CLINICAL TRIAL: NCT00730886
Title: A Randomized Study to Evaluate the Effectiveness and Safety of ExAblate Surgery Compared With Myomectomy for the Enhancement of Fertility Following Treatment of Uterine Fibroids in Women Seeking Pregnancy
Brief Title: ExAblate Treatment of Uterine Fibroids for Fertility Enhancement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: InSightec (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UF023
Record Dates: First submitted 2008-08-05; First posted 2008-08-08 (Estimated); Results first posted 2018-08-15 (Actual); Last update posted 2018-08-15 (Actual); Status verified 2018-08

CONDITIONS: Uterine Fibroids, With Unexplained Infertility
Keywords: Uterine Fibroids; Unexplained Infertility; MRgFUS; ExAblate; Focused Ultrasound; Myomectomy
MeSH Terms: conditions — Leiomyoma | interventions — Uterine Myomectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Non-invasive procedure for fertility enhancement (i.e., ExAblate treatment)
  Interventions: Device: ExAblate 2000
- 2 (Active Comparator): Invasive surgical procedure for fertility enhancement (i.e., myomectomy)
  Interventions: Procedure: Myomectomy

INTERVENTIONS:
Device: ExAblate 2000 — Magnetic resonance image guided focused ultrasound (MRgFUS) for fibroid ablation
  Arms: 1
Procedure: Myomectomy — Invasive surgical procedure for fibroid removal
  Arms: 2

SUMMARY:
The objective of this trial is to evaluate the efficacy and safety of the ExAblate 2000 system for enhancement of fertility in women with non-hysteroscopically resectable uterine fibroids, who are diagnosed with unexplained infertility.

Uterine fibroids are fairly common in women of child-bearing age. An evidence based review supported removing fibroids that distort the uterine cavity to increase pregnancy rates and decrease the rates of miscarriage. Some fibroids can be removed hysteroscopically which is minimally invasive, with low morbidity. However, removal of fibroids within the uterine wall require more invasive surgical procedures (e.g., myomectomy), with increasing morbidity risks including, but not limited to, infection, blood loss and postoperative uterine adhesions.

ExAblate is approved by FDA for the treatment of uterine fibroids; however, its use in patients seeking pregnancy is considered experimental. Accumulated evidence suggests there are no significant complications from the procedure in women seeking pregnancy as with existing fibroid therapies; however, these data are based on a small number of patients. This study will evaluate fertility enhancement following ExAblate treatment or myomectomy, in women with unexplained infertility and who have non-hysteroscopically resectable uterine fibroids.

ELIGIBILITY:
Inclusion Criteria:

Female Partner

1. Able and willing to give consent
2. Able to attend all study visits.
3. At least one fibroid 3.0 cm or larger which is type 2 submucosal or intramural touching or abutting the cavity.
4. Able to communicate sensations during the ExAblate procedure.
5. Uterine fibroids, which are device accessible
6. Fibroids(s) clearly visible on non-contrast MRI. and with uniform enhancement with gadolinium
7. Age 21 to 40 (patients cannot be treated following their 41st birthday)
8. Patients with uterine cavitary distortion based on MRI images or ultrasound.
9. Premenopausal status
10. Normal pap smear and/or HPV testing within institutional guidelines
11. At least one ovary and at least one ipsilateral patent fallopian tube confirmed b hysterosalpingogram or laparoscopy.
12. Normal serum follicle-stimulating hormone and thyrotropin values on days 1-5 of the cycle
13. Length of 2 of the 3 most recent menstrual cycles between 24 and 35 days.
14. History of trying for pregnancy for at least 6 months
15. Documentation of ovulation using urine LH testing, serum LH testing, serum progesterone > 4 ng/dl or endometrial biopsy showing secretory endometrium in a cycle between 24 and 35 days
16. Patient needs to demonstrate that she has already undergone testing and counseling in a fertility clinic or other medical office.

Male partner inclusion criteria

1. Age of male partner < 55
2. At least 10 million total mobile sperm on semen analysis within last 6 months
3. Use of donor sperm which includes at least 10 million total mobile sperm, for female candidates who otherwise meet eligibility criteria (e.g., single women, etc)

Exclusion Criteria:

1. Uterine size > 16 weeks
2. Prior surgical intervention for fibroids (including UAE) except uncomplicated myomectomy (hysteroscopic, laparoscopic or abdominal) and MRgFUS.
3. Prior use of in vitro fertilization or other assisted reproductive technology
4. Previous treatment with gonadotropins or intrauterine inseminations
5. History of tubal surgery
6. History of oophorectomy
7. History of chemotherapy or radiation to the abdomen or pelvis
8. MRI showing only adenomyosis
9. Metallic implants that are incompatible with MRI
10. Severe claustrophobia that would prevent completion of procedure in MR unit
11. Patients with a BMI greater than 38.
12. Known intolerance to the MRI contrast agent (e.g. Gadolinium or Magnevist) including severe kidney disease
13. Individuals who are not able or willing to tolerate the required prolonged stationary prone position during treatment (approximately 3 hrs.)
14. Active pelvic inflammatory disease (PID)
15. Active local or systemic infection
16. Known or suspected pelvic carcinoma or pre-malignant conditions, including sarcoma and adenomatous hyperplasia
17. Dermoid cyst of the ovary anywhere in the treatment path
18. Extensive abdominal scarring that cannot be avoided by redirection of the beam (e.g., due to Caesarean section or repeated abdominal surgeries)
19. Undiagnosed vaginal bleeding
20. Patients having a contraindication to pregnancy.
21. Patients having a contraindication to surgery, including surgical myomectomy
22. Patients with type 0 submucosal fibroids.
23. More than 4 clinically significant fibroids >2cm in mean diameters
24. Patients on dialysis.
25. Hematocrit < 25
26. Hemolytic anemia
27. Patients with unstable cardiac status including:
28. Unstable angina pectoris on medication
29. Patients with documented myocardial infarction within six months of protocol entry
30. Congestive heart failure requiring medication (other than diuretic)
31. Patients on anti-arrhythmic drugs
32. Severe hypertension (diastolic BP > 100 on medication)
33. Patients with cardiac pacemakers
34. Patients planning to use adjuvant therapies post (ExAblate or Myomectomy) procedures to improve the chance of conception within 9 months of study treatment will be excluded from study (note: candidates relying on donor sperm and artificial insemination to conceive between months 3 and 9 post-treatment are allowed to participate, provided they meet all eligibility criteria)
35. Patients without uterine cavity distortion.

Male partner exclusion criteria

1. Prior use of in vitro fertilization of other assisted reproductive technology
2. Previous treatment intrauterine inseminations
3. History of chemotherapy or radiation to the abdomen or pelvis
4. History of vasovasectomy
5. History of varicocelectomy
6. History of pelvic-node dissection
7. Use of calcium-channel blocking medications

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2008-07; Primary Completion 2011-07 (Actual); Study Completion 2011-10-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (6):
- United States (6):
  - UCLA, Los Angeles, California
  - Atlanta Interventional Institute, Smyrna, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - Duke University, Durham, North Carolina
  - Willowbend Health and Wellness, Plano, Texas
  - University of Virginia Health System, Charlottesville, Virginia

REFERENCES:
- [Background] Hanstede MM, Tempany CM, Stewart EA. Focused ultrasound surgery of intramural leiomyomas may facilitate fertility: a case report. Fertil Steril. 2007 Aug;88(2):497.e5-7. doi: 10.1016/j.fertnstert.2006.11.103. Epub 2007 Feb 8. PMID 17292361
- [Background] Rabinovici J, David M, Fukunishi H, Morita Y, Gostout BS, Stewart EA; MRgFUS Study Group. Pregnancy outcome after magnetic resonance-guided focused ultrasound surgery (MRgFUS) for conservative treatment of uterine fibroids. Fertil Steril. 2010 Jan;93(1):199-209. doi: 10.1016/j.fertnstert.2008.10.001. Epub 2008 Nov 14. PMID 19013566
- [Derived] Bouwsma EV, Gorny KR, Hesley GK, Jensen JR, Peterson LG, Stewart EA. Magnetic resonance-guided focused ultrasound surgery for leiomyoma-associated infertility. Fertil Steril. 2011 Jul;96(1):e9-e12. doi: 10.1016/j.fertnstert.2011.04.056. Epub 2011 May 13. PMID 21570071
- See also: Sponsor's Web Page — http://www.insightec.com

RESULTS

PARTICIPANT FLOW:
Groups:
- ExAblate Treatment:: All patients who received at least 10 therepeutic sonications with the ExAblate 2000 Magnetic resonance image guided focused ultrasound (MRgFUS) for fibroid ablation.
- Myomectomy Treatment:: All patients who had more than 15 grams of fibroid tissue excised.
Period: Overall Study
Arm/Group | ExAblate Treatment: | Myomectomy Treatment:
Started | 2 | 0 (no subjects enrolled in this arm. Study enrollment terminated early.)
Completed | 0 | 0 (no subjects enrolled in this arm. Study enrollment terminated early.)
Not Completed | 2 | 0
Not completed — Lost to Follow-up | 1 | 0
Not completed — Physician Decision | 1 | 0

BASELINE CHARACTERISTICS:
Population: Study was terminated due to lack of enrollment
Groups:
- Total: Total of all reporting groups
Arm/Group | ExAblate Treatment: | Myomectomy Treatment: | Total
Number analyzed (Participants) | 2 | 0 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 2 |  | 2
  >=65 years | 0 |  | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 |  | 2
  Male | 0 |  | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 |  | 0
  Asian | 1 |  | 1
  Native Hawaiian or Other Pacific Islander | 0 |  | 0
  Black or African American | 0 |  | 0
  White | 1 |  | 1
  More than one race | 0 |  | 0
  Unknown or Not Reported | 0 |  | 0

OUTCOME MEASURES:

1. Primary Outcome: Live Birth Rate
Time Frame: Between the 3 and 9-month post-treatment visits
Population: enrollment in the clinical trial did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results.
Arm/Group | ExAblate Treatment: | Myomectomy Treatment:
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Pregnancy Rate
Time Frame: Between the 3 and 15-month post-treatment visits
Population: as for outcome 1
Arm/Group | ExAblate Treatment: | Myomectomy Treatment:
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Term Delivery Rate
Time Frame: Between the 3 and 15-month post-treatment visits
Population: as for outcome 1
Arm/Group | ExAblate Treatment: | Myomectomy Treatment:
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Miscarriage Rate
Time Frame: Between the 3 and 15-month post-treatment visits
Population: as for outcome 1
Arm/Group | ExAblate Treatment: | Myomectomy Treatment:
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time to Conception
Time Frame: Post-treatment
Population: as for outcome 1
Arm/Group | ExAblate Treatment: | Myomectomy Treatment:
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: C-Section Rate
Time Frame: Post-treatment
Population: as for outcome 1
Arm/Group | ExAblate Treatment: | Myomectomy Treatment:
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Uterine Fibroid Symptom and Health-Related Quality of Life Questionnaire (UFS-QOL)
Time Frame: Post-treatment
Population: as for outcome 1
Arm/Group | ExAblate Treatment: | Myomectomy Treatment:
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Center for Epidemiologic Studies Depression Scale (CES-D)
Time Frame: Post-treatment
Population: as for outcome 1
Arm/Group | ExAblate Treatment: | Myomectomy Treatment:
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Medical Outcomes Study 36-Item Short Form Survey
Time Frame: Post-treatment
Population: as for outcome 1
Arm/Group | ExAblate Treatment: | Myomectomy Treatment:
Number analyzed (Participants) | 0 | 0

10. Secondary Outcome: Health Care Costs
Time Frame: Post-treatment
Population: as for outcome 1
Arm/Group | ExAblate Treatment: | Myomectomy Treatment:
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | ExAblate Treatment: | Myomectomy Treatment:
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/0
Other Adverse Events (participants affected / at risk) | 1/2 | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ExAblate Treatment: (N=2) | Myomectomy Treatment: (N=0)
perinatal fever (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Subject experienced post delivery fever reported to be unrelated to ExAblate treatment. The fever resulted from prolonged ruptured membranes prior to admission for labor and delivery.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ExAblate Treatment: (N=2) | Myomectomy Treatment: (N=0)
blood tinged mucus peri-rectum (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
enrollment in the clinical trial did not reach the target number of subjects needed to achieve target power and was insufficient to produce statistically reliable results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No